CLINICAL TRIAL: NCT03271502
Title: Effect of Inhalation Anesthesia With Sevoflurane and Total Intravenous Anesthesia With Propofol on Optic Nerve Sheath Diameter in Patients Undergoing Robot-assisted Laparoscopic Prostatectomy
Brief Title: Effect of Anesthesia on Optic Nerve Sheath Diameter in Patients Undergoing Robot-assisted Laparoscopic Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, MD, PhD, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2017-1011
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Anesthesia, Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total intravenous anesthesia (Experimental): Total intravenous anesthesia with propofol and remifentanil
  Interventions: Procedure: Total intravenous anesthesia
- Inhalation anesthesia (Active Comparator): Inhalation anesthesia with sevoflurane and remifentanil
  Interventions: Procedure: Inhalation anesthesia

INTERVENTIONS:
Procedure: Total intravenous anesthesia — Total intravenous anesthesia with propofol and remifentanil
  Arms: Total intravenous anesthesia
Procedure: Inhalation anesthesia — Inhalation anesthesia with sevoflurane and remifentanil
  Arms: Inhalation anesthesia

SUMMARY:
The purpose of this study was to evaluate the difference between the optic nerve sheath diameter measured during total intravenous anesthesia and the optic nerve sheath diameter measured during inhalation anesthesia in patients undergoing robot-assisted laparoscopic prostatectomy.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the difference between the optic nerve sheath diameter measured during total intravenous anesthesia with propofol and remifentanil and the optic nerve sheath diameter measured during inhalation anesthesia with sevoflurane and remifentanil in patients undergoing robot-assisted laparoscopic prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

Patients who have undergone a robot-assisted laparoscopic prostatectomy with a prostate cancer and who are 20 years of age or older and under 80 years of age and who agree to participate in this study.

Exclusion Criteria:

Patients with a history of cerebral hemorrhage or cerebral infarction, Patients < 20 years of age, Patients ≥ 80 years of age, Patients with unexpected hemodynamic instability during surgery, Failure to measure optic nerve sheath diameter.

Ages: 20 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Difference in optic nerve sheath diameter | 60 minutes after pneumoperitoneum and steep Trendelenburg position
  Difference between the optic nerve sheath diameter measured during total intravenous anesthesia and the optic nerve sheath diameter measured during inhalation anesthesia

SECONDARY OUTCOMES:
Difference in optic nerve sheath diameter | 30 minutes after pneumoperitoneum and steep Trendelenburg position
  Difference between the optic nerve sheath diameter measured during total intravenous anesthesia and the optic nerve sheath diameter measured during inhalation anesthesia
Difference in optic nerve sheath diameter | 5 minutes after pneumoperitoneum and steep Trendelenburg position
  Difference between the optic nerve sheath diameter measured during total intravenous anesthesia and the optic nerve sheath diameter measured during inhalation anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kug Kim, MD,PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Yu J, Hong JH, Park JY, Hwang JH, Cho SS, Kim YK. Propofol attenuates the increase of sonographic optic nerve sheath diameter during robot-assisted laparoscopic prostatectomy: a randomized clinical trial. BMC Anesthesiol. 2018 Jun 20;18(1):72. doi: 10.1186/s12871-018-0523-7. PMID 29925316